CLINICAL TRIAL: NCT01020890
Title: A Cross-sectional Study on the Prevalence of GERD in Primary Care Patients With Upper GI Symptoms Using the GERD-Q. The Bulgarian GERD-Q Study
Brief Title: Prevalence of Gastroesophageal Reflux Disease in Primary Care Patients With Upper Gastrointestinal Symptoms
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca
Other Study IDs: NIS-GBG-NEX-2009/1
Record Dates: First submitted 2009-11-25; First posted 2009-11-26 (Estimated); Last update posted 2010-07-12 (Estimated); Status verified 2010-07

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: GERD diagnosis; GERD-Q; GERD patients' characteristics; GERD
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to provide data on the gastroesophageal reflux disease (GERD) prevalence as percentage of patients with upper gastrointestinal (GI) symptoms that are identified with GERD using the Gerd-Q Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients with upper gastrointestinal symptoms

Exclusion Criteria:

* History of oesophageal, gastric or duodenal surgery
* Current treatment with antiinflammatory drugs, including OTC
* Current treatment with proton pump inhibitors ang H2-blockers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 2210 (Actual)
Dates: Start 2009-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- Bulgaria (12):
  - Research Site, Blagoevgrad
  - Research Site, Burgas
  - Research Site, Dobrich
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Varna
  - Research Site, Veliko Tarnovo
  - Research Site, Vratsa
  - Research Site, Yambol